CLINICAL TRIAL: NCT00991224
Title: A Pilot, Open Label, Multi Arm, Single Ctr Study to Evaluate Safety & Tolerability of Escalating Doses of Autologous T Cells Modified With Lentiviral Vectors Expressing High Affinity Gag-specific TCRS in HLA-A02 Patients With HIV
Brief Title: Redirected High Affinity Gag-Specific Autologous T Cells for HIV Gene Therapy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Adaptimmune (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Basic Science
Other Study IDs: 810108
Record Dates: First submitted 2009-10-06; First posted 2009-10-07 (Estimated); Last update posted 2019-10-10 (Actual); Status verified 2017-12

CONDITIONS: HIV Infections
Keywords: HIV; HIV therapeutic vaccine
MeSH Terms: conditions — HIV Infections | interventions — Treatment Interruption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm 1 (Experimental): Subjects who are HIV positive, taking medication to control virus, have an undetectable viral load, CD4 count greater than 450 at the time of enrollment, a CD4 nadir >200 and a recorded historical viral load setpoint, will receive a WT-gag-TCR modified autologous T cells, followed one week later by a 16 week treatment interruption.
  Interventions: Biological: WT-gag-TCR modified T cells; Other: STI or Drug Holiday
- Arm 2 (Experimental): Subjects who are HIV positive, taking medication to control virus, have an undetectable viral load, CD4 count greater than 450 at the time of enrollment, a CD4 nadir >200 and a recorded historical viral load setpoint, will receive a α/6-gag-TCR modified autologous T cells, followed one week later by a 16 week treatment interruption.
  Interventions: Biological: α/6-gag-TCR modified T cells; Other: STI or Drug Holiday
- Arm 3 (Experimental): Subjects who are HIV positive, taking medication to control virus, have an undetectable viral load, CD4 count greater than 450 and a CD4 nadir >200. Subject will undergo an 16 week treatment interruption during which a single infusion of WT-gag-TCR modified autologous T cells at 8 weeks post STI.
  Interventions: Biological: WT-gag-TCR modified T cells; Other: STI or Drug Holiday
- Arm 4 (Experimental): Subjects who are HIV positive, taking medication to control virus, have an undetectable viral load, CD4 count greater than 450 and a CD4 nadir of >200. Subject will undergo a 16-week treatment interruption during which a single infusion of α/6-gag-TCR modified autologous T cells at 8 weeks post STI.
  Interventions: Biological: α/6-gag-TCR modified T cells; Other: STI or Drug Holiday

INTERVENTIONS:
Biological: WT-gag-TCR modified T cells — Single dose of WT-gag-TCR modified T cells infused over 3 consecutive days.
  Arms: Arm 1; Arm 3
Biological: α/6-gag-TCR modified T cells — Single dose of WT-gag-TCR modified T cells infused over 3 consecutive days.
  Arms: Arm 2; Arm 4
Other: STI or Drug Holiday — Subjects will stop taking antiviral medications for 16 weeks.

SUMMARY:
This research study is being carried out to study a new way to possibly treat HIV. T-cells are one of the white blood cells used by the body to fight HIV. CD8 T-cells are a type of T-cell used by the body to detect and kill cells which have been infected by foreign viruses or organisms, including the HIV virus. CD8 T-cells must identify the HIV virus in order to kill it. Because HIV is constantly changing the way it looks to the CD8 T-cells, some of the HIV virus escapes detection and is not killed by the CD8 T-cells.

This research study uses a T cell receptor (TCR) protein specific for HIV (SL9 TCR) and adds it to the CD8 T-cells in the laboratory in order to help the CD8 T-cells recognize the constantly changing HIV virus and make it able to fight HIV more efficiently. TCR stands for T cell receptor. TCRs are found on the surface of T cells and allow the T cells to recognize other cells. Laboratory studies have shown that when CD8 T-cells are modified with SL9 TCRs, they kill cells that are infected with HIV better than normal CD8 T-cells can. On the basis of these laboratory results, there is the potential that SL9 TCRs may work in people infected with HIV and improve their immune system by killing HIV infected cells and thus may help control HIV infection.

Two different SL9 TCRs will be tested in this study, WT-gag-TCR and α/6-gag-TCR. Two different types of SL9 TCRs are being used in this research study because the laboratory studies suggest that the different SL9 TCRs will function differently depending on the amount of virus in your body. A goal of this clinical study is to test the effects of infusions of either SL9 TCR in the presence or absence of a viral load.

All subjects who receive WT-gag-TCR or the α/6-gag-TCR T cells will be enrolled in a Long Term Follow up study to monitor subjects. Subjects will be followed every 6 months for five years following the 1st infusion of the T cells. If the WT-gag-TCR or the α/6-gag-TCR T cells are no longer found in the blood after five years, then subjects will be contacted yearly for the next 10 years. If the WT-gag-TCR or the α/6-gag-TCR T cells are found in the blood at five years after the 1st infusion of T cells, then the subjects will continue to be seen once a year until the WT-gag-TCR or the α/6-gag-TCR T cells are no longer found in the blood for a maximum of 15 years.

DETAILED DESCRIPTION:
See Above

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Karnofsky Performance of 80 or higher
* HLA-A2 Positive
* Chronic HIV-1 infection
* On stable HAART regimen (with no changes within 4 weeks of study entry)
* Willing to undergo a limited treatment interruption of antiretroviral medication
* CD4+ T cell count ≥450 cells/mm3
* Documented CD4 nadir of ≥200 cells/mm3
* Undetectable HIV-1 RNA
* ARMS 1 and 2 only, at least a singe documented historic viral load set point reading
* Lab Values: Hgb≥10 males; ≥9.5 females ; ANC≥1000/mm3 ; Platelets≥1000,000/mm3 ; Creatinine≤1.5 mg/dL ; AST, ALT ≤ 2.5xULN

Exclusion Criteria:

* Current or prior AIDS diagnosis
* Previous participation in any gene therapy using an integrating vector (subjects treated with Placebo will not be excluded)
* History of cancer or malignancy (allowed to have successfully treated basal cell or squamous cell carcinoma of the skin)
* Have history or current exam indicative of active or unstable cardiac disease or hemodynamic instability
* Have history or current exam indicative of bleeding diathesis
* Previous treatment with any HIV experimental vaccine within 6 months prior to screening
* Use of chronic corticosteroids, hydroxyurea or immunomodulating agents such as IL2, interferon alpha, interferon gamma, granulocyte colony stimulating factors within 30 days prior to study entry (inhaled steroids are not exclusionary)
* Currently breast feeding, pregnant or unwilling to use acceptable methods of birth control
* Use of aspirin, dipyridamole, warfarin or any other medication that is likely to affect platelet function or other aspects of blood coagulation during the 2 week period prior to leukapheresis
* Active drug or alcohol use/dependence
* Serious illness requiring systemic treatment and/or hospitalization within 30 days prior to study entry
* Receipt of a vaccination within 30 days prior to study entry
* Have a known allergy or hypersensitivity to human serum albumin, DMSO or Dextran 40

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-11; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
To determine optimal dose and to evaluate the safety and tolerability of the study drug. | 3 years from end of study
To monitor for delayed adverse events associated with lentiviral vector gene transfer (RCL and insertional oncogenesis) | 3 years from end of study

SECONDARY OUTCOMES:
To determine the antiviral effects of WT-gag-and α/6-gag- TCR transduced cells in patients with low and high antigen load (presence and absence of viremia) | 3 years from end of study
To monitor engraftment of vector modified cells in the peripheral circulation | 3 years from end of study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: UPenn AIDS Clinical Trials Unit (ACTU) Website — http://www.uphs.upenn.edu/pennactu/